CLINICAL TRIAL: NCT02485431
Title: A Single-Dose, Single-Center, Randomized, Five Period Crossover Study Comparing Food Effect and Bioavailability of Deflazacort Formulations in Healthy Volunteers
Brief Title: Food Effect and Bioavailability of Deflazacort Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Collaborators: ICON Development Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MP-104-CL-026
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Deflazacort, fasted (Experimental): 36mg of Deflazacort with 240 ml of room-temperature, non-carbonated water in Fasted state.
  Interventions: Drug: Deflazacort
- Deflazacort, high-fat meal (Experimental): 36mg of Deflazacort with 240 ml of room-temperature, non-carbonated water with high fat meal served 30 minutes prior to dosing.
  Interventions: Drug: Deflazacort
- Deflazacort, crushed, fasted (Experimental): 36mg of Deflazacort crushed and mixed with apple sauce.
  Interventions: Drug: Deflazacort
- Deflazacort alternate strength,fasted (Experimental): Investigational Formulation Deflazacort tablet (6 X 6mg).
  Interventions: Drug: Deflazacort
- Deflazacort suspension with apple juice (Experimental): Deflazacort oral suspension (36mg) mixed with 100ml apple juice in fasted state.
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort
  Other Names: DFZ

SUMMARY:
This is a Phase 1, single-center, single-dose, randomized, 5-period crossover study designed to assess the comparative bioavailability and food effect of deflazacort. A total of 45 subjects will be randomly assigned to receive 1 of 5 treatment sequences. Each dosing sequence will be enrolled in parallel and all subjects will receive all 5 treatments in a crossover fashion.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, single-dose, randomized, 5-period crossover study designed to assess the comparative bioavailability and food effect of deflazacort. A total of 45 subjects will be randomly assigned to 1 of 5 treatment sequences. Each dosing sequence will be enrolled in parallel and will receive all 5 treatments in a crossover fashion.

Subjects will be screened within 28 days of the first dose of study drug. Subjects will check into the clinical pharmacology unit (CPU) on the day prior to dosing (Day -1 for Period 1) and will stay in-house through the 24 hour assessments in each study period. Safety assessments will be performed at screening, check-in for each period, and at 24 hours after each dose per the Schedule of Assessments .Additionally, a safety follow-up phone call will be performed on Day 36 (± 2 days).

Subject participation is expected to last approximately 64 days, including a 28-day screening period and a 36-day on study period (consisting of 5 treatment periods, washout periods lasting 7 days, and the safety follow-up phone call).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥ 18 and ≤ 55 at the time of screening.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2, inclusive, at screening and Day -1.
* Women of nonchildbearing potential, defined as tubal ligation, hysterectomy, postmenopausal (amenorrhea for > 1 year; confirmed by FSH), or oophorectomy.
* Males who are sexually active and whose partners are females of childbearing potential must agree to use condoms from screening through 90 days after the last dose of study drug.
* Males must agree to not donate sperm from screening through 90 days after the last dose of study drug.
* Subjects must be healthy and without clinically significant abnormalities as assessed by review of medical and surgical history, physical examination, vital signs measurement, electrocardiogram (ECG), and laboratory evaluations conducted at the screening visit and on CPU admission.
* Subjects must be nonsmokers, defined as having abstained from tobacco- or nicotine-containing products (eg, cigarettes, chewing tobacco, snuff, nicotine patches, and electronic cigarettes) in the 3 months prior to screening.

Exclusion Criteria:

* Positive pregnancy test or lactating.
* History or presence of conditions which, in the judgment of the investigator, are known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History or presence of conditions that may place the subject at increased risk as determined by the investigator.
* History of presence of hypersensitivity of idiosyncratic reaction to the study drugs or related compounds (eg, steroids or their formulations including lactose).
* History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of screening.
* Use of prescription medications within 14 days or any drugs that inhibit study drug specific cytochrome P450(s) within 14 days or any drugs that induce specific cytochrome P450s, including St. John's Wort, within 28 days, or 5 half-lives, whichever is longer, of administration of the first dose of study drug and throughout the study.
* Use of over the-counter (OTC) drugs (including herbal preparations) within 7 days or 5 half-lives, whichever is longer, prior to administration of the first dose of study drug and throughout the study.
* Has taken other investigational drugs, including deflazacort or related compounds, or participated in any clinical study within 30 days or 5 half-lives of the investigational drug's PK, pharmacodynamic, or biological activity, whichever is longer, prior to first dose of study drug in this study.
* Has received any immunosuppressive agents, coal tar, and/or radiation therapies within 30 days prior to the first dose of study drug.
* Has received injectable corticoids in the 12 weeks prior to the first dose of study drug or any oral form of corticoids in the 30 days prior to the first dose of study drug.
* Has received any live or live-attenuated vaccine within 30 days prior to the first dose of study drug and/or intends to receive one on study.
* Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
* Positive urine drugs of abuse, alcohol breath test, or urine cotinine screen.
* Positive screen for human immunodeficiency virus (HIV)-1 and HIV-2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
* Estimated creatinine clearance < 80 mL/min using Cockcroft-Gault equation.
* QTcF interval > 450 msec at screening.
* Unwilling or unable to consume standardized meals.
* Unwilling or unlikely to comply with the requirements of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile | Day 30
  Pharmacokinetic parameters such as the maximum observed plasma concentration (Cmax), time to Cmax (Tmax), the area under the plasma concentration versus time curve from time 0 (predose) to the last quantifiable time point (AUClast), AUC from time 0 (predose) to time infinity (AUCinf), the elimination rate constant (λz), and terminal elimination half-life (t½) will be calculated

SECONDARY OUTCOMES:
Treatment emergent AEs and SAEs | Day 30
  Incident of treatment -emergent AEs (TEAEs) and SAEs
Changes from baseline values for lab | Day 30
  Changes from baseline values for clinical laboratory test.
Changes from baseline values for ECG | Day 30
  Changes from baseline values for ECG
Changes from baseline values for physical exam | Day 30
  Changes from baseline values for physical exam
Changes from baseline values for vital signs | Day 30
  Changes from baseline values for vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Uma Arumugam, MD, Study Director — ICON Development Solutions, LLC
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States